CLINICAL TRIAL: NCT05161195
Title: A Post-trial Access Roll-over Study to Allow Access to Ribociclib (LEE011) for Patients Who Are on Ribociclib Treatment in Novartis-sponsored Study
Brief Title: Roll-over Study to Allow Continued Access to Ribociclib
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011A2412B; 2024-514891-41-00 (Registry Identifier: EU CT Number)
Expanded Access: NCT05038631 (Available)
Record Dates: First submitted 2021-12-03; First posted 2021-12-17 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer
Keywords: Roll-over Protocol; Post Trial Access (PTA); Ribociclib (LEE011); Ribociclib in combination with other drugs; Hormone Receptor (HR); HR-positive; Human Epidermal Growth Factor Receptor 2 (HER2); HER2-negative; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Letrozole; Anastrozole; Goserelin; Tamoxifen; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ribociclib (Other): Participants will receive ribociclib with other drugs at the same dose and schedule as in the parent study. Treatment continues until clinical benefit ends (e.g., disease progression), unacceptable toxicity, consent withdrawal, protocol non-compliance, transition to alternative therapy or access program, can receive ribociclib through prescription (commercially availability and reimbursement of ribociclib except for U.S. participants from CLEE011A2404).
  Interventions: Drug: Ribociclib; Drug: Letrozole; Drug: Anastrozole; Drug: Goserelin; Drug: Tamoxifen; Drug: Fulvestrant

INTERVENTIONS:
Drug: Ribociclib — Participants continue ribociclib as was administered in their parent study
  Other Names: LEE011
Drug: Letrozole — Participants continue ribociclib in combination with letrozole as was administered in their parent study
Drug: Anastrozole — Participants continue ribociclib in combination with anastrozole as was administered in their parent study
Drug: Goserelin — Participants continue ribociclib in combination with goserelin as was administered in their parent study
Drug: Tamoxifen — Participants continue ribociclib in combination with tamoxifen as was administered in their parent study
Drug: Fulvestrant — All participants continue ribociclib in combination with fulvestrant as was administered in their parent study

SUMMARY:
The purpose of this study is to assess the long-term safety of ribociclib (LEE011) in combination with other drugs and provide post-trial access (PTA) to participants who are currently receiving treatment with ribociclib in combination with other drugs and continuing to have clinical benefit in a Novartis-sponsored global study that has reached its primary objective(s).

DETAILED DESCRIPTION:
This is an open-label, multi-center, roll-over study to evaluate the long-term safety of ribociclib in combination with other drugs in participants who are participating in a Novartis sponsored global study, that has fulfilled requirements for its primary objective(s), and who in the opinion of the Investigator, would benefit from continued treatment.

This roll-over study will not include a screening phase, participants will directly transfer at the completion of the parent study. Eligible participants will start receiving ribociclib in combination with other drugs (as per parent protocol) only after they have signed the Informed Consent and have met the selection criteria for this roll-over study.

Participants should return to the study center for resupply of the study medication and for safety and clinical benefit assessment, at a minimum, every 24 weeks, or more frequently at any given time required as per local practice.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Participant is currently participating in a Novartis sponsored global study (parent study), receiving treatment with ribociclib in combination with other drugs and the parent study has fulfilled its primary objective(s).
* Willingness and ability to comply with scheduled visits, treatment plans and any other study procedures.
* Participant must have been receiving treatment with ribociclib for at least 6 cycles in the parent study.
* Participant must have evidence of clinical benefit as determined by the Investigator.

Key Exclusion Criteria:

* Permanent discontinuation of ribociclib in the parent study due to toxicity or disease progression, non-compliance to study procedures, withdrawal of consent or any other reason as stipulated in parent protocol.
* Participant currently has unresolved toxicities for which ribociclib dosing has been interrupted in the parent study (participants meeting all other eligibility criteria may be enrolled once toxicities have resolved to allow ribociclib dosing to resume).
* Local access to commercially available ribociclib and reimbursed (except for US enrolled participants from parent protocol CLEE011A2404 meeting all other eligibility criteria).
* Women of child-bearing potential defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during the study treatment and for 21 days after stopping the treatment. Highly effective contraception methods include:

  1. Total abstinence
  2. Female sterilization
  3. Male partner sterilization
  4. Placement of an intrauterine device (IUD)
* Male contraception during ribociclib use by male participants is not required unless it is necessary due to the safety profile of other medications a participant is taking or by local regulations.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2030-06-28 (Estimated); Study Completion 2030-08-14 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with treatment-emergent adverse events (AES) | From day of first dose of study medication to 30 days after last dose of study medication, up to 8 years
  The percentage of participants with treatment-emergent adverse events will be summarized, including significant adverse events leading to discontinuation, and adverse events leading to dose adjustment

SECONDARY OUTCOMES:
Clinical benefit rate | Up to 8 years
  Percentage of participants with clinical benefit as assessed by the Investigator at scheduled study visits

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (67):
- United States (16):
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mid Florida Hematology And Onc Ctr, Orange, Florida
  - Summit Cancer Care, Savannah, Georgia
  - John D Archbold Memorial Hospital, Thomasville, Georgia
  - Duly Health and Care, Plainfield, Illinois
  - Indian Univ Health Goshen Center forCancer, Goshen, Indiana
  - Northern Light Mercy Hospital, Portland, Maine
  - Englewood Health, Englewood, New Jersey
  - The Valley Hospital-Luckow Pavillion, Paramus, New Jersey
  - Eastchester Center for Cancer Care, The Bronx, New York
  - University Hospitals of Cleveland Seidman Cancer Center, Cleveland, Ohio
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - Millennium Research Clin Develop, Houston, Texas
- Novartis Investigative Site, San Juan, Argentina
- Brazil (6):
  - Novartis Investigative Site, Natal, Rio Grande do Norte
  - Novartis Investigative Site, Ijuí, Rio Grande do Sul
  - Novartis Investigative Site, Florianópolis, Santa Catarina
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Sao Jose Rio Preto
  - Novartis Investigative Site, São Paulo
- China (13):
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Kunming, Yunnan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Qingdao
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Novartis Investigative Site, San José, Costa Rica
- Novartis Investigative Site, Heraklion Crete., Greece
- Novartis Investigative Site, Hong Kong, Hong Kong
- India (2):
  - Novartis Investigative Site, Bhubaneshwar, Odisha
  - Novartis Investigative Site, Delhi
- Novartis Investigative Site, Meldola, FC, Italy
- Japan (3):
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Koto Ku, Tokyo
- Lebanon (2):
  - Novartis Investigative Site, El Chouf, LBN
  - Novartis Investigative Site, Beirut
- Novartis Investigative Site, San Pedro G G, Mexico
- Peru (2):
  - Novartis Investigative Site, Trujillo, La Libertad
  - Novartis Investigative Site, San Borja, Lima region
- Novartis Investigative Site, Gdansk, Poland
- Portugal (3):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Loures
  - Novartis Investigative Site, Porto
- Novartis Investigative Site, Singapore, Singapore
- South Africa (3):
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Johannesburg
  - Novartis Investigative Site, Pretoria
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Novartis Investigative Site, Sant Joan Despí, Barcelona, Spain
- Novartis Investigative Site, Taipei, Taiwan
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Malatya, Battalgazi
  - Novartis Investigative Site, Diyarbakır, Sur
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kecioren Ankara
- Novartis Investigative Site, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com